CLINICAL TRIAL: NCT00110851
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of the Effects of PN2034 in Type 2 Diabetes Patients on Concomitant Rosiglitazone and Metformin (or Avandamet) Therapy
Brief Title: Safety and Efficacy Study of PN2034 in Type 2 Diabetes Patients on Concomitant Rosiglitazone and Metformin (or Avandamet)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wellstat Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PN2034.05.001
Record Dates: First submitted 2005-05-13; First posted 2005-05-16 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes, type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone; Metformin

INTERVENTIONS:
Drug: rosiglitazone
Drug: metformin
Drug: PN2034

SUMMARY:
This study is designed to evaluate the safety and efficacy of PN2034 administered to type 2 diabetics on concomitant rosiglitazone and metformin (or Avandamet) therapy as measured by change in glycosylated hemoglobin (HbA1c) levels from baseline to Week 12. Also the study will evaluate the effect of PN2034 on glucose control as measured by fasting plasma glucose (FPG) and on fasting lipid levels: triglycerides, total cholesterol, high-density lipoproteins (HDL), low-density lipoproteins (LDL), and very low-density lipoproteins (VLDL).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 2 diabetes mellitus
* 21 to 72 years of age
* taking rosiglitazone and metformin (or Avandamet) for at least 3 months, and on a stable dose of rosiglitazone (or Avandamet) for at least 2 months
* glycosylated hemoglobin (HbA1c) level of >/=7.5% but </=10.0%
* fasting blood sugar level >/= 125 mg/dL but </= 279 mg/dL
* BMI 26-43 kg/m2
* direct bilirubin < 1.5x the upper limit of normal (ULN)
* serum creatinine < 1.5 mg/dL (males) or < 1.4 mg/dL (females)
* blood urea nitrogen (BUN)</=40 mg/dL
* all other clinical laboratory parameters (hematology, serum chemistry, and urinalysis) within normal limits or not clinically significant
* ECG normal, or abnormalities not clinically significant
* surgically sterile, postmenopausal, or using adequate contraception and have a negative pregnancy test at Screening
* willing and able to sign an informed consent form

Exclusion Criteria:

* diagnosed with type 1 diabetes mellitus or has a history of ketoacidosis
* treatment with insulin, TZDs (excluding rosiglitazone) or any other oral or injected antidiabetic (excluding metformin or Avandamet) within 3 months prior to screening or during study treatment
* change in lipid-lowering medication within 2 months of screening
* taken systemic corticosteroids within 1 month prior to screening or during study treatment
* history of or current/active cardiovascular disease
* significant current pulmonary conditions
* significant thyroid disease
* CPK value > 3x ULN
* a female who is pregnant or lactating
* systolic BP > 160 mm Hg or a diastolic BP > 90 mm Hg at screening
* previous or current history of cancer, other than basal cell or stage 1 squamous cell carcinoma of the skin, that has not been in remission within 5 years prior to randomization
* liver function tests (ALT, AST, ALP) > 2 times ULN, or active liver disease at screening
* history of positive HIV
* positive hepatitis B test at screening
* weight loss or gain >/= 15 lbs within 3 months of screening
* history of substance abuse (including alcohol abuse) within 2 years prior to screening
* donated and/or received any blood or blood products within 3 months prior to randomization
* taken an investigational study medication within 30 days prior to screening or during the study

Ages: 21 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2005-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety
Effect on HbA1c levels

SECONDARY OUTCOMES:
Effect on glucose control as measured by FPG
Effect on lipid levels

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Phoenix Internal Medicine Associates, Waterbury, Connecticut
  - University Clinical Research-DeLand, DeLand, Florida
  - Center for Diabetes and Endocrine Care, Hollywood, Florida
  - Genesis Research International, Longwood, Florida
  - Baptist Diabetes Associates, Miami, Florida
  - Andres Patron, DO PA, Pembroke Pines, Florida
  - CLIRECO, Inc., Tamarac, Florida
  - Endocrine Clinical Research, Winter Park, Florida
  - PRN of Kansas, Wichita, Kansas
  - Medical Research Associates of Charlotte, Charlotte, North Carolina
  - Neem Research Group of Charlotte, Charlotte, North Carolina
  - Unifour Medical Research Associates, Hickory, North Carolina
  - Neem Research Group of Raleigh, Raleigh, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Camp Hill Clinical Research Center, Camp Hill, Pennsylvania
  - Neem Research Group, Columbia, South Carolina
  - Palmetto Medical Research Associates, Mt. Pleasant, South Carolina
  - Oaks Medical Center, Spring, Texas